CLINICAL TRIAL: NCT01133119
Title: Use of Local Anesthetic (0.25% Bupivacaine) for Pain Control in Pediatric Cardiac Catheterization: A Randomized Controlled Trial.
Brief Title: Use of Local Anesthetic (0.25% Bupivacaine) for Pain Control in Pediatric Cardiac Catheterization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lee Benson, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000013970
Record Dates: First submitted 2010-04-01; First posted 2010-05-28 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2013-08

CONDITIONS: Pain
Keywords: cardiac catheterization; local anesthetic; pain experienced post-operatively; pediatric patients
MeSH Terms: conditions — Pain | interventions — Standard of Care; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Active Comparator)
  Interventions: Drug: Standard of Care
- Treatment Group 2 (Experimental)
  Interventions: Drug: Standard of Care plus bupivacaine

INTERVENTIONS:
Drug: Standard of Care — Subjects will have femoral sheaths removed under general anesthetic but without subcutaneous infiltration of bupivacaine.
  Arms: Treatment Group 1
Drug: Standard of Care plus bupivacaine — Subcutaneous dose of 0.25% bupivacaine infiltrated around the entry site of the femoral artery/vein sheath, just prior to sheath removal.
  Participants will receive a dose of up to 0.8mL/kg (up to 2.0 mg/kg) of 0.25% bupivacaine, with the final amount at the discretion of the physician.
  Arms: Treatment Group 2

SUMMARY:
In the Cardiac Diagnostic and Interventional Unit (CDIU) at the Hospital for Sick Children (SickKids), minimally invasive procedures are performed to diagnose and treat a variety of congenital heart defects. Procedures are performed under general anesthetic and involve inserting a catheter through the skin and into the femoral vein or artery in the groin. In addition, the use of local anesthetic as a pain control regimen just prior to the removal of femoral artery or vein sheaths is used by some but not all cardiac interventionalists. Local anesthetic is infiltrated near the sheath insertion site, at the end of the procedure while the child is under general anesthetic, with the goal of decreasing pain at the insertion site and promoting comfort in the post-operative period. The use of local anesthetic depends on the choice of the individual practitioner and is not currently a routine practice for all patients.

The investigators proposed research seeks to investigate whether the use of subcutaneous bupivacaine reduces pain levels in the post-operative period in children having cardiac catheterization procedures.

DETAILED DESCRIPTION:
A number of differences in pediatric cardiac catheterization procedures exist that limit the transferability of research findings from the adult literature. For example, the majority of pediatric cardiac catheterizations are performed under general anesthetic, and femoral sheaths are removed while under general anesthetic and at the end of the procedure. In contrast in adult clinical practice, procedures are not performed under general anesthetic, and femoral sheaths are removed when patients are awake and often 4 to 6 hours after the end of the procedure. These differences limit the ability to apply research findings in adults to pediatrics, warranting further study of the effects of local anesthetic on femoral site pain in children. As well, studies in adults have examined pain only up to 20 minutes after sheath removal. We seek to investigate the impact of bupivacaine up to 6 hours after cardiac catheterization in children.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 7-18 years
2. Scheduled for cardiac catheterization through the femoral artery and/or vein under general anesthetic
3. Ability to speak and understand English
4. No apparent cognitive impairments

Exclusion Criteria:

1. Known allergies to bupivacaine
2. Impaired renal function
3. Impaired hepatic function

Ages: 7 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Self-reported levels of pain | For 6 hours after admission to the CDIU
  The primary outcome measure is self-reported levels of pain using the Numerical Rating Scale (NRS). Patients will be asked to verbally rate the amount of femoral pain experienced between 0-10 on admission to CDIU recovery, and at 15 and 30 minutes, and 1, 2, 4, and 6 hours after admission.
  We will be examining the change in pain scores over time as well as the total pain experienced by the paitents. These measures will be compared between the two treatment groups.

SECONDARY OUTCOMES:
Use of analgesics | 6 hours post-operatively
  Intervention groups will be able to receive additional analgesia as needed, and the type and amount of medication received will be recorded by nursing staff
Use of a suture to close the femoral artery | Post-operatively
  If used, this suture is removed post-operatively and may influence post-operative pain levels. We would like to record whether a suture was used and removed as part of our data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Benson, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: Link to published study results — http://onlinelibrary.wiley.com/doi/10.1002/ccd.26284/epdf